CLINICAL TRIAL: NCT04514549
Title: Assessing Emerald and MC10 nPoint Biosensors for Rett Syndrome
Brief Title: ASSESSING EMERALD AND MC10 BIOSTAMP nPOINT BIOSENSORS FOR RETT SYNDROME
Status: Completed | Type: Observational
Sponsor: Rett Syndrome Research Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SENS-101-RSRT
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Rett Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: will enroll approximately 5 patients with pronounced respiratory dysfunction. Patients may be enrolled with tremors and or seizures. All patients will be observed via Emerald to capture sleep staging, movement and breathing for up to approximately 4 weeks. Caregivers will keep a daily questionnaire diary of the patient's anxiety, sleep and seizures. MC10 nPoint data will be captured for at least two 24-hour periods in each of the 4 weeks to assess patch placements for breathing detection. Ongoing assessment of MC10 nPoint data may lead to the use of more or less sensors, changes in duration of sensor data collection, or placement as Cohort 1 progresses.Preliminary results from Cohort 1 will determine if Emerald will continue to be evaluated and will inform on MC10 nPoint optimizations for Cohort 2. If preliminary results indicate Emerald is not an effective device, then Emerald will be discontinued
  Interventions: Device: Emerald
- Cohort 2: will enroll approximately 15 patients. Patients with pronounced respiratory dysfunction, tremors, seizures, and/or other expanded features of Rett syndrome deemed appropriate may be enrolled. If Emerald is continued, all patients are observed via Emerald to capture sleep staging, movement and breathing up to for approximately 4 weeks. Caregivers will keep a daily questionnaire diary of the patient's anxiety, sleep and seizures. Ongoing assessment of MC10 nPoint data may lead to the use of more or less sensors, changes in duration of sensor data collection, or placement as Cohort 2 progresses.

INTERVENTIONS:
Device: Emerald — The Emerald is a wireless sensor that can track the motion, breathing, and sleep of subjects without touching or requiring any interaction with the subjects, allowing them to go about their normal lives. The physical device is roughly a 30 x 35 x 5 cm box that contains directional antennas and a motherboard to process these signals. In typical operation, the device is mounted onto a wall within a clinic or home setting using peel-away (reversible) mount strips.
  Other Names: MC 10
  Groups: Cohort 1

SUMMARY:
This is a pilot study of the Emerald device in Rett syndrome patients diagnosed with a confirmed MECP2 mutation. MC10 BioStamp nPoint patches will also be assessed with the goal to develop Rett-specific breathing algorithms

DETAILED DESCRIPTION:
The study consists of two sequential cohorts with a total of approximately 20 patients enrolled. Patients in each cohort may participate for up to 4 weeks. Each participant will have up to 2 Emerald devices installed in their home for monitoring sleep, breathing and movement, and will use between 3 and 9 nPoint patches for determining proper patch placement for detecting breathing signals.

The study will consist of a Screening visit, an Observation period, and a Follow-up phone call. The Screening Period will be one day in clinic, the Observation period will be up to 4 weeks at home and the Follow up phone call will be performed at the completion of the Observation Period.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to the conduct of any study-specific procedures, the parent/caregiver/LAR must provide written informed consent. If the caregiver attending the clinic visits is not the parent or LAR, written consent must be obtained from the parent or LAR for the caregiver's participation in the study.
2. Diagnosis of typical Rett Syndrome according to the revised Clinical Diagnostic Criteria1 and presence of a disease causing MECP2 genetic mutation.
3. The patient's parent/caregiver/LAR must be able to understand the nature of the study and to allow for the completion of study assessments. The same parent/caregiver/LAR must be capable of providing reliable information about the patient's condition.
4. Live within approximately 50 to 60 miles of MIT.
5. Primary language English.
6. Approximately 4 people or less living in the home. This does not include visiting caregivers.
7. Must have home access to Wi-Fi.

Exclusion Criteria:

1. Inability of patient to sleep alone in their own room.
2. Pets in the home, or caregivers unwilling to keep pets out of the bedroom monitored by Emerald during the Observation Period.
3. Plans to take a prolonged vacation or to otherwise be out of the home during the Observation Period.
4. Participation in another device study that could interfere with this study.
5. Active implantable devices such as pacemakers or defibrillators.
6. Known allergies or hypersensitivities to adhesives.
7. Patients with any condition that, in the opinion of the principal investigator, might interfere with the conduct of the study, confound interpretation of the study results, endanger their own well-being, or who may otherwise not be suitable for the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female patients with Diagnosis of typical Rett Syndrome according to the revised Clinical Diagnostic Criteria and presence of a disease-causing MECP2 genetic mutation.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Emerald respiratory function in Rett patients | 4 weeks
  Suitability of Emerald technology to assess sleep staging and

SECONDARY OUTCOMES:
MC10 | 8 weeks
  Determination of MC10 BioStamp nPoint patch placement for detecting breathing

CONTACTS AND LOCATIONS:
Overall Officials: David Lieberman, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No